CLINICAL TRIAL: NCT01973426
Title: Development and Evaluation of a Human-Machine Interface for Grasp Assistance Using a Robotic Thumb Orthosis in Children With Hemiplegic Cerebral Palsy and Hemiplegic Stroke
Brief Title: Evaluating Human-Machine Interfaces in a Robotic Thumb Orthosis
Acronym: IOTA
Status: Completed | Type: Observational
Sponsor: Wyss Institute at Harvard University (Other)
Collaborators: Boston Children's Hospital (Other); Deborah Munroe Noonan Memorial Research Fund (Other)
Responsible Party: Sponsor
Other Study IDs: AMD-CS-0026
Record Dates: First submitted 2013-10-24; First posted 2013-10-31 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Hemiplegic Stroke; Hemiplegic Cerebral Palsy
Keywords: Robot; Thumb; Orthosis; Hemiplegia; Hemiplegic Stroke; Hemiplegic Cerebral Palsy; Stroke; Cerebral Palsy; Grasp assistance
MeSH Terms: conditions — Hemiplegia; Stroke; Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with limited control of their thumb: Children afflicted by hemiplegic stroke or hemiplegic cerebral palsy who have lost the ability to actively (and accurately) control the thumb.
  Interventions: Device: Isolated Orthosis for Thumb Actuation (IOTA)

INTERVENTIONS:
Device: Isolated Orthosis for Thumb Actuation (IOTA) — In this pilot study, we plan to investigate whether the IOTA can effectively facilitate the ability of participants to perform a specific set of clinically relevant tasks conducted in a clinic setting. The IOTA is a device developed at the Wyss Institute at Harvard University, in collaboration with Children's Hospital Boston, for assisting opposable thumb grasping tasks. The IOTA contains an adjustable brace fitted to the thumb and dorsum of the hand that is easy to put on and facilitates grasping motions through flexible cable-driven actuators that assist with joint abduction and extension.

SUMMARY:
We plan to investigate whether the Isolated Orthosis for Thumb Actuation (IOTA) can effectively facilitate the ability of participants to perform a specific set of clinically relevant tasks conducted in a clinic setting.

DETAILED DESCRIPTION:
Many Activities of Daily Living involve precision grasp and fine motor manipulation, such as putting toothpaste on a toothbrush or feeding oneself. However, children afflicted by stroke, cerebral palsy, or traumatic brain injury may lose the ability to actively (and accurately) control the thumb, and specifically abduct/adduct the carpometacarpal (CMC) joint and flex/extend the metacarpophalangeal (MCP) joint. We are testing the Isolated Orthosis for Thumb Actuation (IOTA), a device developed at the Wyss Institute at Harvard University in collaboration with Children's Hospital Boston, for assisting opposable thumb grasping tasks. The IOTA contains an adjustable brace fitted to the thumb and dorsum of the hand that is easy to put on and facilitates grasping motions through flexible cable-driven actuators that assist with CMC joint abduction and MCP joint extension.

In this pilot study, we plan to investigate whether the IOTA can effectively facilitate the ability of participants to perform a specific set of clinically relevant tasks conducted in a clinic setting.

The hypothesis for this work is that the IOTA will significantly improve the participant's performance on clinically relevant tasks.

ELIGIBILITY:
Inclusion Criteria:

* Be between 7 - 16 years old
* Have a clinical diagnosis of hemiplegic cerebral palsy or hemiplegic stroke causing a thumb contracture affecting one hand
* Not have a diagnosis of dystonia
* Have completed at least a 6-week post-operative period following hand surgery (if applicable; self-reported)
* Be able to follow instructions (as determined by their attending Occupational Therapist)
* Not be allergic to nylon or lycra

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with hemiplegic cerebral palsy or hemiplegic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Investigate whether the IOTA can effectively facilitate a participant's ability to perform a specific set of clinically relevant tasks in a clinical setting. | 1 study session per participant, lasting up to 2 hours.
  We will examine this aim by evaluating participant performance on a Box and Block Task. This task is clinically relevant to the participant population. This task will be evaluated with no device worn at first, and then with the IOTA device worn in four different modes (manual mode, cycle & repeat mode, wrist mode, and moon mode).

CONTACTS AND LOCATIONS:
Overall Officials: Leia Stirling, Ph.D., Principal Investigator — Wyss Institute at Harvard University; Annette Correia, OT, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States